CLINICAL TRIAL: NCT05119647
Title: The Efficacy and Safety Study of Thrombus Aspiration Catheter(Ton-bridgeMT) on Endovascular Treatment of Acute Ischemic Stroke
Brief Title: A Single-Arm Objective Performance Criteria Trial for Intracranial Thrombus Aspiration Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ton-Bridge Medical Tech. Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZHTQ2021001
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke; Aspiration; Catheter; Intracranial
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Aspiration thrombectomy (Experimental): Since this is a single-arm objective performance criteria trial, patients with acute stoke caused by artery occlusion shall not be divided into two groups.
  Interventions: Device: Thrombus Aspiration Catheter(Ton-bridgeMT)

INTERVENTIONS:
Device: Thrombus Aspiration Catheter(Ton-bridgeMT) — Thrombus Aspiration Catheter is a developed technique for treating acute stroke caused by artery occlusion. The catheter(Ton-bridgeMT) was specially designed for those patients who experience acute stroke within 24 hours.

SUMMARY:
This is a prospective multicenter, single-arm objective performance criteria trial to assess the efficacy and safety of the the thrombus aspiration catheter.

DETAILED DESCRIPTION:
The study is conducted in 15 centers all around China, aiming at recruiting 155 patients with acute stroke caused by artery occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Baseline NIHSS score ≥6;
* Subject has acute occlusion located in Vertebral artery(VA) / Internal Carotid Artery (ICA) / M1or M2 segment of Middle Cerebral Artery (MCA) / Basilar artery (BA) diagnosed by DSA;
* Femoral artery puncture is expected to be completed within 24 hours of onset；
* mRS score≤ 2;
* Subject or legal representative is able to understand the purpose of study, agrees to comply with protocol requirements and has provided written informed consent.

Exclusion Criteria:

* Chronic occlusion in the target area;
* Epilepsy at the time of stroke；
* Bleeding from the gastrointestinal or urinary system in the past three weeks；
* After drug control, systolic blood pressure was greater than 185mmhg and / or diastolic blood pressure was greater than 110mmhg;
* International Normalized Ratio(INR)>3;
* Random blood glucose < 2.7mmol/L or > 22.2mmol/L;
* Heart, lung, liver, kidney failure or other serious diseases (such as brain tumors, - systemic infection, active disseminated intravascular coagulation, myocardial infarction within 12 months before enrollment, history of severe mental illness);
* Tortuous lesion / severe stenosis in the starting segment of the carotid artery / Carotid dissection / Arteritis judged by researchers that is not suitable for the procedure;
* Acute occlusion of bilateral carotid arteries；
* Intracranial hemorrhage or massive infarction diagnosed by CT or MR;
* History of allergies to antiplatelet drugs, anticoagulants, anesthetics, contrast agents;
* Expected life <12 months;
* Female subjects who are pregnant or planning to become pregnant or lactate within the study period;
* Subject has participated in any other drug or medical device clinical trials in 1 month before signing informed consent;
* Other circumstances judged by researchers that are not suitable for enrollment .

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Successful recanalization rate within three-times aspiration | Up to 90 days
  Successful recanalization is defined as modified Thrombolysis In Cerebral Infarction scale(mTICI) 2b or 3 evaluated by Digital subtraction angiography (DSA).

SECONDARY OUTCOMES:
Successful recanalization rate within three-times aspiration | Intraoperation
  Successful recanalization is defined as mTICI 2b or 3 evaluated by DSA.
Successful recanalization rate beyond three-times aspiration | Intraoperation
  Successful recanalization is defined as mTICI 2b or 3 evaluated by DSA. Auxiliary device such as stent could be used.
National Institute of Health stroke scale(NIHSS) | 72 hours / 7 days
  NIHSS score in 72 hours and 7 days(or the day when patients discharged, depends on which day is earlier) will be compared.
Rate of Modified Rankin Scale(mRS) score less than 3 | 90 days
  The mRS score is assessed in 90 days follow-up.
Device delivery performance | Intraoperation
  Device delivery performance including transport and pullback performance, which is ranked excellent/good/normal/bad.
The rate of symptomatic intracranial hemorrhage | 72 hours
  National Institute of Health stroke scale(NIHSS) increased by at least 4 compared with the baseline.
Death rate | Up to 90 days
  Subjects who died from any cause would be counted.
The rate of AE | Up to 90 days
  The definition of AE(Adverse Event) refers to ISO 14155
The rate of SAE | Up to 90 days
  The definition of SAE (Serious Adverse Event) refers to ISO 14155
The rate of medical device deficiency | Up to 90 days
  Medical device deficiency refer to the unreasonable risks of medical devices that may endanger human health and life safety under normal use in the process of clinical trials, such as label errors, quality problems, malfunctions, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Liqun Jiao, Principal Investigator — Xuanwu Hospital, Beijing
Locations (15):
- China (15):
  - The First Affiliated Hospital of USTC, Hefei, Anhui
  - Zhuhai people's hospital, Zhuhai, Guangdong
  - The Second Nanning People's hospital, Nanning, Guangxi
  - Cangzhou central hospital, Cangzhou, Hebei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Ganzhou Municipal Hospital, Ganzhou, Jiangxi
  - Central Hospital Affiliated to Shangdong First Medical University, Jinan, Shandong
  - First People's Hospital of Jinan, Jinan, Shandong
  - The Second People's Hospital of Liaocheng, Liaocheng, Shandong
  - Rizhao central Hospital, Rizhao, Shandong
  - Shanxi Candiovascular hospital, Taiyuan, Shanxi
  - School of medicine UESTC, Chengdu, Sichuan
  - Zigong Third People's Hospital, Zigong, Sichuan
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Xuanwu hospital Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: No